CLINICAL TRIAL: NCT04969484
Title: Improving Palliative Care Access Through Technology (ImPAcTT): A Multi- Component Pilot Study
Brief Title: Improving Palliative Care Access Through Technology
Acronym: ImPAcTT
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: K76 grant transferred to new institution (NOA 3/2020). COVID-19 significantly impacted study team personnel & study setting; human subjects restrictions at both the University and CMS levels prevented any human subjects research for more than a year.
Sponsor: University of Utah (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Caroline Stephens, PhD, RN, GNP-BC, FAAN, Helen Lowe Bamberger Colby Presidential Endowed Chair in Gerontological Nursing, Associate Professor, University of Utah
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB_00129094; 5K76AG054862-05 (NIH)
Record Dates: First submitted 2021-05-04; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Telehealth; Palliative Care
Keywords: End of life; Care transition; Nursing Home
MeSH Terms: conditions — Death

STUDY DESIGN:
Intervention Model Description: The trial will be implemented in 3 nursing homes to evaluate the feasibility and acceptability of the multi-component ImPAcTT intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ImPAcTT intervention (Experimental): Within 48-72 hours of enrollment in the study, the primary participant and family will receive an ImPAcTT Telehealth visit with the PC provider. The provider will conduct a comprehensive PC assessment aligned with the National Consensus Project for Quality Palliative Care guidelines. Visits, which may include remote physical assessment using a digital stethoscope, dermatoscope, etc., will be documented and transmitted to the NH. Advanced Care Planning (ACP) and goals of care discussions will be facilitated by the ability to virtually share and edit documents, such as the Physician Orders for Life Sustaining Treatment (POLST), in real time with primary participants and/or family. The PC provider will conduct follow-up visits 1 week following the initial visit, then on a case-by-case basis.
  Interventions: Other: Telehealth visit
- Usual care (No Intervention): Participants will receive the standard of care established at the NH.

INTERVENTIONS:
Other: Telehealth visit — ImPACTT Telehealth visit with the PC provider
  Arms: ImPAcTT intervention

SUMMARY:
This project will focus on developing, optimizing and pilot-testing a multi-component Improving Access Through Technology (ImPAcTT) intervention that leverages existing telehealth technologies to provide staff education; family outreach, engagement and support; care coordination; and resident symptom management and facilitation of goals-of-care discussion.

DETAILED DESCRIPTION:
Almost 1.8 million older Americans live in nursing homes (NH), with estimates that this number will grow to more than 3 million by 2050. NHs are increasingly becoming the place of care and site of death for frail older adults dying from multiple chronic illnesses. Unfortunately, most residents die without the benefit of palliative care (PC) or with palliation delayed until the last days of life.

Unfortunately, hospice services are often the only formal end of life care service available in NHs, and access to hospice enrollment is complicated by financial implications for both NHs and residents.

Telehealth, or remote monitoring of patients through information and communication technologies, is an effective mechanism for addressing the increased demand on health services and has much to offer to people living with and dying from advanced illness. Moreover, numerous studies have demonstrated positive benefits of using telehealth in the NH to improve access to consultants (e.g., neurology, dermatology, psychiatry).

Little is known, however, about the effect of using Telehealth on improving access to PC specialists in the NH setting.

The proposed ImPAcTT intervention employs a secure communications platform that permits multi-person live video, audio, and text message consultations; real-time document sharing and documentation for advanced care planning discussions; and remote virtual assessment capabilities.

The investigator will conduct a pilot implementation trial of ImPAcTT in 3 study nursing homes to evaluate our ability to safely recruit and retain study participants, collect appropriate and accurate data, and determine preliminary estimates of an effect size of the intervention.

ELIGIBILITY:
Purposeful sampling will take place in an attempt to collect data from a range of ethnically and racially diverse participants.

INCLUSION CRITERIA:

Primary participant

* Age >= 18 years
* English language fluency
* Palliative Care Consult Screening Tool (PCCS) scoring 9 or above
* If participant does not demonstrate capacity to consent, he/she must be able to assent to study procedures, be told of plan to approach surrogate and have a legally authorized representative available to provide consent

Family/friend caregivers:

* Closest relative/next of kin/friend who is involved in the care of his/her loved one before and during the study period
* English fluency

EXCLUSION CRITERIA:

Primary participant:

* Enrolled in hospice
* Unable to assent to study procedures
* Expresses resistance or dissent to participation or the use of surrogate consent

Family/friend caregiver:

* Life expectancy < 1 year (e.g., metastatic cancer)
* Evidence of cognitive impairment or inability to consent to study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2018-02-19 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Symptom distress (composite measure) | Baseline and Last visit -12 weeks
  Symptom distress as measured by the Edmonton Symptom Assessment Scale - ESAS
  * ESAS physical score (total of physical 6 symptoms, score range 0-60)
  * ESAS emotional score (total of 2 emotional symptoms, score range 0-60)
  * ESAS total symptom distress score (physical score + emotional score + well being)
  For all symptom distress scores:
  High score means: worst outcome Low score means: better outcome
Change in Symptom impact | Baseline and Last visit -12 weeks
  Symptom impact as measured by the "Quality of Life at the End of Life" - QUAL-E
  Symptom impact subscale:
  Minimum value: 3 Maximum value: 15
  High score means: worst outcome Low score means: better outcome

SECONDARY OUTCOMES:
Change in number of completed POLST forms | Baseline and Last visit -12 weeks
  Number of Physician's Orders for Life-Sustaining Treatment - POLST forms completed
Type of changes in POLST forms | Baseline and Last visit -12 weeks
  Type of changes in Physician's Orders for Life-Sustaining Treatment -POLST forms
Number of In-hospital death | Baseline and Last visit -12 weeks
  Number of In-hospital death
Change in Family Satisfaction | Baseline and Last visit -12 weeks
  Family Satisfaction as measured by the "Quality of Life at the End of Life - Family" - QUAL-E Fam
  Subscale: Relationship with Healthcare Provider [Questions #5-8 with 5 item Likert scales, average of 4 scores] Minimum value: 1 Maximum value: 5
  High score means: worst outcome Low score means: better outcome
Number of residents transitioned to hospice | Last visit - week 12
  Number of residents transitioned to hospice
Change in acute care utilization (composite measure) | Baseline and Last visit -12 weeks
  Number of ED Visits and number of Hospitalizations
Change in Functional Status | Baseline and Last visit -12 weeks
  Functional Status as measured by the PalliativePerformance Scale (PPSv2)
  Minimum value: 0% Maximum value: 100%
  High score means: better outcome Low score means: worst outcome
Change in Depression Status | Baseline and Last visit -12 weeks
  Depression as measured by the Patient Health Questionnaire-9 (PHQ-9)
  Subscales:
  - Question 1: Minimum value: 0 Maximum value: 27
  High score means: worst outcome Low score means: better outcome
  - Question 2: Minimum value: 1 Maximum value: 4
  High score means: worst outcome Low score means: better outcome
Change in Cognitive Status | Baseline and Last visit -12 weeks
  Cognition as measured by the Montreal - Cognitive Assessment (MoCA)
  Minimum value: 0 Maximum value: 30
  High score means: better outcome Low score means: worst outcome
Change in Mortality | Baseline and Last visit -12 weeks
  Risk for dying within one year as measured by the Flacker Mortality Score
  Minimum value: 0 Maximum value: 15.21
  High score means: worst outcome Low score means: better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Caroline E Stephens, PhD, RN, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - University of California San Francisco - UCSF, San Francisco, California
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Data (complete dataset with full documentation including metadata, protocols, etc) will be made available by the online publication date unless the NIH policy specifies an earlier date. The PI will work the primary mentor to ensure that the study data are submitted to the PCRC De-identified Data Repository. (https://palliativecareresearch.org/corescenters/data-informatics-statistics-core-disc/pcrc-de-identified-data-repository-didr).
  This would allow for secondary data analyses of the data to be conducted and support those who need access to these datasets for preliminary data and/or grant proposal preparation. Human subject data will be shared with other investigators within the limits of HIPAA and other patient confidentiality requirements, including the removal of all participant identifiers from all source documents and the use of unique participant identification numbers, and in accordance with PCRC protocols.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available by the online publication date unless the NIH policy specifies an earlier date.
Access Criteria: This study has specific data and resource sharing plans to make data available both to the community of scientists interested in palliative care and nursing home research to avoid unintentional duplication of research. Moreover, the investigator would welcome collaboration with others who could make use of the Telehealth visit protocols developed in this ImPAcTT project.
URL: https://palliativecareresearch.org/corescenters/data-informatics-statistics-core-disc/pcrc-de-identified-data-repository-didr

REFERENCES:
- [Result] Mitchell SL, Teno JM, Miller SC, Mor V. A national study of the location of death for older persons with dementia. J Am Geriatr Soc. 2005 Feb;53(2):299-305. doi: 10.1111/j.1532-5415.2005.53118.x. PMID 15673356
- [Result] National Center for Health Statistics (US). Health, United States, 2010: With Special Feature on Death and Dying. Hyattsville (MD): National Center for Health Statistics (US); 2011 Feb. Report No.: 2011-1232. Available from http://www.ncbi.nlm.nih.gov/books/NBK54381/ PMID 21634072
- [Result] Brock DB, Foley DJ. Demography and epidemiology of dying in the U.S. with emphasis on deaths of older persons. Hosp J. 1998;13(1-2):49-60. doi: 10.1080/0742-969x.1998.11882887. PMID 9644392
- [Result] Bercovitz A, Decker FH, Jones A, Remsburg RE. End-of-life care in nursing homes: 2004 National Nursing Home Survey. Natl Health Stat Report. 2008 Oct 8;(9):1-23. PMID 19013934
- [Result] Kaye HS, Harrington C, LaPlante MP. Long-term care: who gets it, who provides it, who pays, and how much? Health Aff (Millwood). 2010 Jan-Feb;29(1):11-21. doi: 10.1377/hlthaff.2009.0535. PMID 20048355
- [Result] Stephens C, Halifax E, Bui N, Lee SJ, Harrington C, Shim J, Ritchie C. Provider Perspectives on the Influence of Family on Nursing Home Resident Transfers to the Emergency Department: Crises at the End of Life. Curr Gerontol Geriatr Res. 2015;2015:893062. doi: 10.1155/2015/893062. Epub 2015 Aug 24. PMID 26379704
- [Result] Stephens CE, Halifax E, David D, Bui N, Lee SJ, Shim J, Ritchie CS. "They Don't Trust Us": The Influence of Perceptions of Inadequate Nursing Home Care on Emergency Department Transfers and the Potential Role for Telehealth. Clin Nurs Res. 2020 Mar;29(3):157-168. doi: 10.1177/1054773819835015. Epub 2019 Apr 21. PMID 31007055
- [Result] Gozalo P, Teno JM, Mitchell SL, Skinner J, Bynum J, Tyler D, Mor V. End-of-life transitions among nursing home residents with cognitive issues. N Engl J Med. 2011 Sep 29;365(13):1212-21. doi: 10.1056/NEJMsa1100347. PMID 21991894
- [Result] Miller SC, Lima JC, Looze J, Mitchell SL. Dying in U.S. nursing homes with advanced dementia: how does health care use differ for residents with, versus without, end-of-life Medicare skilled nursing facility care? J Palliat Med. 2012 Jan;15(1):43-50. doi: 10.1089/jpm.2011.0210. Epub 2011 Dec 16. PMID 22175816
- [Result] Cohen A, Bulanda JR. Social Supports as Enabling Factors in Nursing Home Admissions: Rural, Suburban, and Urban Differences. J Appl Gerontol. 2016 Jul;35(7):721-43. doi: 10.1177/0733464814566677. Epub 2015 Jan 11. PMID 25582118
- [Result] Bolin JN, Phillips CD, Hawes C. Urban and rural differences in end-of-life pain and treatment status on admission to a nursing facility. Am J Hosp Palliat Care. 2006 Jan-Feb;23(1):51-7. doi: 10.1177/104990910602300109. PMID 16450663
- [Result] Douthit N, Kiv S, Dwolatzky T, Biswas S. Exposing some important barriers to health care access in the rural USA. Public Health. 2015 Jun;129(6):611-20. doi: 10.1016/j.puhe.2015.04.001. Epub 2015 May 27. PMID 26025176
- [Result] Matthews KA, Croft JB, Liu Y, Lu H, Kanny D, Wheaton AG, Cunningham TJ, Khan LK, Caraballo RS, Holt JB, Eke PI, Giles WH. Health-Related Behaviors by Urban-Rural County Classification - United States, 2013. MMWR Surveill Summ. 2017 Feb 3;66(5):1-8. doi: 10.15585/mmwr.ss6605a1. PMID 28151923
- [Result] Aragon K, Covinsky K, Miao Y, Boscardin WJ, Flint L, Smith AK. Use of the Medicare posthospitalization skilled nursing benefit in the last 6 months of life. Arch Intern Med. 2012 Nov 12;172(20):1573-9. doi: 10.1001/archinternmed.2012.4451. PMID 23026981
- [Result] Ersek M, Carpenter JG. Geriatric palliative care in long-term care settings with a focus on nursing homes. J Palliat Med. 2013 Oct;16(10):1180-7. doi: 10.1089/jpm.2013.9474. Epub 2013 Aug 28. PMID 23984636
- [Result] Casarett D, Pickard A, Bailey FA, Ritchie C, Furman C, Rosenfeld K, Shreve S, Chen Z, Shea JA. Do palliative consultations improve patient outcomes? J Am Geriatr Soc. 2008 Apr;56(4):593-9. doi: 10.1111/j.1532-5415.2007.01610.x. Epub 2008 Jan 16. PMID 18205757
- [Result] Finlay IG, Higginson IJ, Goodwin DM, Cook AM, Edwards AG, Hood K, Douglas HR, Normand CE. Palliative care in hospital, hospice, at home: results from a systematic review. Ann Oncol. 2002;13 Suppl 4:257-64. doi: 10.1093/annonc/mdf668. No abstract available. PMID 12401699
- [Result] Hall S, Kolliakou A, Petkova H, Froggatt K, Higginson IJ. Interventions for improving palliative care for older people living in nursing care homes. Cochrane Database Syst Rev. 2011 Mar 16;2011(3):CD007132. doi: 10.1002/14651858.CD007132.pub2. PMID 21412898
- [Result] Berkowitz RE, Jones RN, Rieder R, Bryan M, Schreiber R, Verney S, Paasche-Orlow MK. Improving disposition outcomes for patients in a geriatric skilled nursing facility. J Am Geriatr Soc. 2011 Jun;59(6):1130-6. doi: 10.1111/j.1532-5415.2011.03417.x. Epub 2011 Jun 7. PMID 21649622
- [Result] Miller SC, Dahal R, Lima JC, Intrator O, Martin E, Bull J, Hanson LC. Palliative Care Consultations in Nursing Homes and End-of-Life Hospitalizations. J Pain Symptom Manage. 2016 Dec;52(6):878-883. doi: 10.1016/j.jpainsymman.2016.05.017. Epub 2016 Sep 17. PMID 27650008
- [Result] Miller SC, Lima JC, Intrator O, Martin E, Bull J, Hanson LC. Palliative Care Consultations in Nursing Homes and Reductions in Acute Care Use and Potentially Burdensome End-of-Life Transitions. J Am Geriatr Soc. 2016 Nov;64(11):2280-2287. doi: 10.1111/jgs.14469. Epub 2016 Sep 19. PMID 27641157
- [Result] Stephens CE, Hunt LJ, Bui N, Halifax E, Ritchie CS, Lee SJ. Palliative Care Eligibility, Symptom Burden, and Quality-of-Life Ratings in Nursing Home Residents. JAMA Intern Med. 2018 Jan 1;178(1):141-142. doi: 10.1001/jamainternmed.2017.6299. PMID 29159368
- [Result] Casarett D, Karlawish J, Morales K, Crowley R, Mirsch T, Asch DA. Improving the use of hospice services in nursing homes: a randomized controlled trial. JAMA. 2005 Jul 13;294(2):211-7. doi: 10.1001/jama.294.2.211. PMID 16014595
- [Result] Zerzan J, Stearns S, Hanson L. Access to palliative care and hospice in nursing homes. JAMA. 2000 Nov 15;284(19):2489-94. doi: 10.1001/jama.284.19.2489. PMID 11074779
- [Result] Happ MB, Capezuti E, Strumpf NE, Wagner L, Cunningham S, Evans L, Maislin G. Advance care planning and end-of-life care for hospitalized nursing home residents. J Am Geriatr Soc. 2002 May;50(5):829-35. doi: 10.1046/j.1532-5415.2002.50207.x. PMID 12028168
- [Result] Johnston B, Kidd L, Wengstrom Y, Kearney N. An evaluation of the use of Telehealth within palliative care settings across Scotland. Palliat Med. 2012 Mar;26(2):152-61. doi: 10.1177/0269216311398698. Epub 2011 Mar 4. PMID 21378067
- [Result] Low JA, Beins G, Lee KK, Koh E. Last moments of life: can telemedicine play a role? Palliat Support Care. 2013 Aug;11(4):353-5. doi: 10.1017/S1478951512000995. Epub 2013 Feb 7. PMID 23388081
- [Result] Wowchuk SM, McClement S, Bond J Jr. The challenge of providing palliative care in the nursing home part II: internal factors. Int J Palliat Nurs. 2007 Jul;13(7):345-50. doi: 10.12968/ijpn.2007.13.7.24346. PMID 17851378
- [Result] Travis SS, Loving G, McClanahan L, Bernard M. Hospitalization patterns and palliation in the last year of life among residents in long-term care. Gerontologist. 2001 Apr;41(2):153-60. doi: 10.1093/geront/41.2.153. PMID 11327480
- [Result] Teno JM, Branco KJ, Mor V, Phillips CD, Hawes C, Morris J, Fries BE. Changes in advance care planning in nursing homes before and after the patient Self-Determination Act: report of a 10-state survey. J Am Geriatr Soc. 1997 Aug;45(8):939-44. doi: 10.1111/j.1532-5415.1997.tb02963.x. PMID 9256845
- [Result] Teno JM, Clarridge BR, Casey V, Welch LC, Wetle T, Shield R, Mor V. Family perspectives on end-of-life care at the last place of care. JAMA. 2004 Jan 7;291(1):88-93. doi: 10.1001/jama.291.1.88. PMID 14709580
- [Result] Miller SC, Teno JM, Mor V. Hospice and palliative care in nursing homes. Clin Geriatr Med. 2004 Nov;20(4):717-34, vii. doi: 10.1016/j.cger.2004.07.005. PMID 15541622
- [Result] Huskamp HA, Stevenson DG, Chernew ME, Newhouse JP. A new medicare end-of-life benefit for nursing home residents. Health Aff (Millwood). 2010 Jan-Feb;29(1):130-5. doi: 10.1377/hlthaff.2009.0523. PMID 20048371
- [Result] Stevenson DG, Bramson JS. Hospice care in the nursing home setting: a review of the literature. J Pain Symptom Manage. 2009 Sep;38(3):440-51. doi: 10.1016/j.jpainsymman.2009.05.006. PMID 19735904
- [Result] Ding J, Saunders C, Cook A, Johnson CE. End-of-life care in rural general practice: how best to support commitment and meet challenges? BMC Palliat Care. 2019 Jun 25;18(1):51. doi: 10.1186/s12904-019-0435-4. PMID 31238934
- [Result] Carlson MD, Lim B, Meier DE. Strategies and innovative models for delivering palliative care in nursing homes. J Am Med Dir Assoc. 2011 Feb;12(2):91-8. doi: 10.1016/j.jamda.2010.07.016. Epub 2010 Nov 10. PMID 21266284
- [Result] Lupu D; American Academy of Hospice and Palliative Medicine Workforce Task Force. Estimate of current hospice and palliative medicine physician workforce shortage. J Pain Symptom Manage. 2010 Dec;40(6):899-911. doi: 10.1016/j.jpainsymman.2010.07.004. PMID 21145468
- [Result] Edirippulige S, Martin-Khan M, Beattie E, Smith AC, Gray LC. A systematic review of telemedicine services for residents in long term care facilities. J Telemed Telecare. 2013 Apr;19(3):127-132. doi: 10.1177/1357633X13483256. Epub 2013 May 23. PMID 23612520
- [Result] Rogante M, Giacomozzi C, Grigioni M, Kairy D. Telemedicine in palliative care: a review of systematic reviews. Ann Ist Super Sanita. 2016 Jul-Sep;52(3):434-442. doi: 10.4415/ANN_16_03_16. PMID 27698303
- [Result] Oliver DP, Demiris G, Wittenberg-Lyles E, Washington K, Day T, Novak H. A systematic review of the evidence base for telehospice. Telemed J E Health. 2012 Jan-Feb;18(1):38-47. doi: 10.1089/tmj.2011.0061. Epub 2011 Nov 15. PMID 22085114
- [Result] Capurro D, Ganzinger M, Perez-Lu J, Knaup P. Effectiveness of eHealth interventions and information needs in palliative care: a systematic literature review. J Med Internet Res. 2014 Mar 7;16(3):e72. doi: 10.2196/jmir.2812. PMID 24610324
- [Result] Kidd L, Cayless S, Johnston B, Wengstrom Y. Telehealth in palliative care in the UK: a review of the evidence. J Telemed Telecare. 2010;16(7):394-402. doi: 10.1258/jtt.2010.091108. Epub 2010 Sep 2. PMID 20813893
- [Result] McCall K, Keen J, Farrer K, Maguire R, McCann L, Johnston B, McGill M, Sage M, Kearney N. Perceptions of the use of a remote monitoring system in patients receiving palliative care at home. Int J Palliat Nurs. 2008 Sep;14(9):426-31. doi: 10.12968/ijpn.2008.14.9.31121. PMID 19060793
- [Result] Roglieri JL, Futterman R, McDonough KL, Malya G, Karwath KR, Bowman D, Skelly J, Warburton SW Jr. Disease management interventions to improve outcomes in congestive heart failure. Am J Manag Care. 1997 Dec;3(12):1831-9. PMID 10178473
- [Result] Lind L, Karlsson D. A system for symptom assessment in advanced palliative home healthcare using digital pens. Med Inform Internet Med. 2004 Sep-Dec;29(3-4):199-210. doi: 10.1080/14639230400005966. PMID 15742987
- [Result] Mair F, Whitten P. Systematic review of studies of patient satisfaction with telemedicine. BMJ. 2000 Jun 3;320(7248):1517-20. doi: 10.1136/bmj.320.7248.1517. PMID 10834899
- [Result] Hammett L, Harvath TA, Flaherty-Robb M, Sawyer G, Olson D. Remote wound care consultation for nursing homes: using a web-based assessment and care planning tool. J Gerontol Nurs. 2007 Nov;33(11):27-35; quiz 36-7. doi: 10.3928/00989134-20071101-09. PMID 18019116
- [Result] Rabinowitz T, Murphy KM, Amour JL, Ricci MA, Caputo MP, Newhouse PA. Benefits of a telepsychiatry consultation service for rural nursing home residents. Telemed J E Health. 2010 Jan-Feb;16(1):34-40. doi: 10.1089/tmj.2009.0088. PMID 20070161
- [Result] Yeung A, Johnson DP, Trinh NH, Weng WC, Kvedar J, Fava M. Feasibility and effectiveness of telepsychiatry services for chinese immigrants in a nursing home. Telemed J E Health. 2009 May;15(4):336-41. doi: 10.1089/tmj.2008.0138. PMID 19441951
- [Result] Biglan KM, Voss TS, Deuel LM, Miller D, Eason S, Fagnano M, George BP, Appler A, Polanowicz J, Viti L, Smith S, Joseph A, Dorsey ER. Telemedicine for the care of nursing home residents with Parkinson's disease. Mov Disord. 2009 May 15;24(7):1073-6. doi: 10.1002/mds.22498. PMID 19353687
- [Result] Michener L, Cook J, Ahmed SM, Yonas MA, Coyne-Beasley T, Aguilar-Gaxiola S. Aligning the goals of community-engaged research: why and how academic health centers can successfully engage with communities to improve health. Acad Med. 2012 Mar;87(3):285-91. doi: 10.1097/ACM.0b013e3182441680. PMID 22373619
- [Result] Frank L, Basch E, Selby JV; Patient-Centered Outcomes Research Institute. The PCORI perspective on patient-centered outcomes research. JAMA. 2014 Oct 15;312(15):1513-4. doi: 10.1001/jama.2014.11100. No abstract available. PMID 25167382
- [Result] Collier A, Morgan DD, Swetenham K, To TH, Currow DC, Tieman JJ. Implementation of a pilot telehealth programme in community palliative care: A qualitative study of clinicians' perspectives. Palliat Med. 2016 Apr;30(4):409-17. doi: 10.1177/0269216315600113. Epub 2015 Aug 19. PMID 26290500
- [Result] May C, Harrison R, Finch T, MacFarlane A, Mair F, Wallace P; Telemedicine Adoption Study Group. Understanding the normalization of telemedicine services through qualitative evaluation. J Am Med Inform Assoc. 2003 Nov-Dec;10(6):596-604. doi: 10.1197/jamia.M1145. Epub 2003 Aug 4. PMID 12925553
- [Result] Yellowlees PM. Successfully developing a telemedicine system. J Telemed Telecare. 2005;11(7):331-5. doi: 10.1258/135763305774472024. PMID 16238833
- [Result] Miller EA. Solving the disjuncture between research and practice: telehealth trends in the 21st century. Health Policy. 2007 Jul;82(2):133-41. doi: 10.1016/j.healthpol.2006.09.011. Epub 2006 Oct 13. PMID 17046097
- [Result] Stillman D, Strumpf N, Capezuti E, Tuch H. Staff perceptions concerning barriers and facilitators to end-of-life care in the nursing home. Geriatr Nurs. 2005 Jul-Aug;26(4):259-64. doi: 10.1016/j.gerinurse.2005.06.002. PMID 16109300
- [Result] Froggatt K. Evaluating a palliative care education project in nursing homes. Int J Palliat Nurs. 2000 Mar;6(3):140-6. doi: 10.12968/ijpn.2000.6.3.8941. PMID 11051950
- [Result] Ouslander JG, Bonner A, Herndon L, Shutes J. The Interventions to Reduce Acute Care Transfers (INTERACT) quality improvement program: an overview for medical directors and primary care clinicians in long term care. J Am Med Dir Assoc. 2014 Mar;15(3):162-170. doi: 10.1016/j.jamda.2013.12.005. PMID 24513226
- [Result] Levy C, Morris M, Kramer A. Improving end-of-life outcomes in nursing homes by targeting residents at high-risk of mortality for palliative care: program description and evaluation. J Palliat Med. 2008 Mar;11(2):217-25. doi: 10.1089/jpm.2007.0147. PMID 18333736
- [Result] Saliba D, Buchanan J, Edelen MO, Streim J, Ouslander J, Berlowitz D, Chodosh J. MDS 3.0: brief interview for mental status. J Am Med Dir Assoc. 2012 Sep;13(7):611-7. doi: 10.1016/j.jamda.2012.06.004. Epub 2012 Jul 15. PMID 22796362
- [Result] Sandelowski M. What's in a name? Qualitative description revisited. Res Nurs Health. 2010 Feb;33(1):77-84. doi: 10.1002/nur.20362. PMID 20014004
- [Result] Steinhauser KE, Clipp EC, Bosworth HB, McNeilly M, Christakis NA, Voils CI, Tulsky JA. Measuring quality of life at the end of life: validation of the QUAL-E. Palliat Support Care. 2004 Mar;2(1):3-14. doi: 10.1017/s1478951504040027. PMID 16594230
- [Result] Hussey MA, Hughes JP. Design and analysis of stepped wedge cluster randomized trials. Contemp Clin Trials. 2007 Feb;28(2):182-91. doi: 10.1016/j.cct.2006.05.007. Epub 2006 Jul 7. PMID 16829207
- See also: Improving palliative care in nursing homes [online report]. New York: Center to Advance Palliative Care. 2008. — https://www.capc.org/capc-reports-and-publications/
- See also: Corbin J, Strauss A, Strauss AL. Basics of qualitative research. Sage; 2014. — https://us.sagepub.com/en-us/nam/basics-of-qualitative-research/book235578